CLINICAL TRIAL: NCT04885868
Title: Patient Acceptability of the Use of an Autonomous Telephone System for the Delivery of Clinical Follow-up Conversations After Cataract Surgery
Brief Title: Patient Acceptability of Autonomous Telemedicine
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ufonia (Industry)
Collaborators: Buckinghamshire Healthcare NHS Trust (Other); Innovate UK (Other Government)
Responsible Party: Sponsor
Other Study IDs: RXQ
Record Dates: First submitted 2021-04-29; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Cataract After
MeSH Terms: conditions — Capsule Opacification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This study assess acceptability of autonomous conversation as part of cataract surgery follow up. — This study assess acceptability of autonomous conversation as part of cataract surgery follow up.

SUMMARY:
Patients will have an automated call supervised by a human clinician to check how they are after uncomplicated cataract surgery as part of their standard of care. The study aims to evaluate the acceptability of this system through a net promoter score and for a subsection of patients using a qualitative interview.

DETAILED DESCRIPTION:
The study will be a qualitative cohort design. The target will be to recruit 1000 patients who meet the inclusion criteria and provide consent following the process set out below. This represents recruiting 75% of the total projected number of patients who will undergo cataract surgery during the trial period.

Currently at Buckinghamshire Healthcare NHS Trust patients who have uncomplicated cataract surgery are given post-op instructions and assessed for their suitability to undergo telephone follow-up by the nursing team in the discharge lounge. If deemed suitable for a telephone call (equivalent to the criteria for inclusion in this study, including the capacity to consent) a date to expect a telephone follow-up call is given. During the study these patients will also be given an information leaflet and information relating to the study by the nursing team.

The post-op telephone call occurs three weeks later and at the start of this call patients will be asked if they consent to take part as well as if they have any further questions. If they agree to participate in the study their follow-up will be conducted by the autonomous human supervised system as well as additional questions to determine the acceptability of the system. If they decline to participate or are unable to consent (for example, the unlikely event that their capacity has become impaired following surgery), they will have their follow-up conducted by a human clinician as per the current standard of care.

For those patients who provide consent the autonomous human supervised system comprises several conversational elements which occur in order:

1. Greeting and introduction
2. Identification of patient
3. Cataract follow-up symptom questions
4. Patient's queries and frequently asked questions
5. Acceptability questions
6. Closure of call

If all of the questions aren't asked by the autonomous system or the human supervisor feels additional information is required they can ask these at the end of the call. The patient may withdraw from the automated call at any point.

Up to 50 patients (5% of total recruited) who consent to participate will be invited to take part in a subsequent structured telephone interview with a researcher to explore in greater depth their experience of using the system. The interview will last no more that 30 minutes and will be conducted within one week of the follow-up call.

Anonymised data from the patient ratings will undergo standard statistical analysis. The qualitative responses to the reasons why they gave their score as well as the answers to the in-depth interviews will undergo thematic analysis to understand patients' perceptions of having the follow-up conducted by the autonomous human supervised system.

ELIGIBILITY:
Inclusion Criteria:

* Routine, first or second eye cataract surgery with intraocular lens implantation without complications.
* Above the age of 16.
* Capacity to give consent
* Access to a phone number.
* Satisfactory command of English for a phone-based consultation.

Exclusion Criteria:

* Combined glaucoma surgery
* Retinal or glaucoma laser treatment
* Corneal dystrophy or grafts
* Combined vitreoretinal surgery

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing uncomplicated cataract surgery who are suitable for telephone follow up
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-05-24 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
A score out of 10 rating the autonomous system | It is anticipated the study will occur over 3 months
  The patient will score the autonomous system out of 10 and a subsection of patients will have qualitative interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Mole, BSc MBBS MSc, Principal Investigator — Ufonia

IPD SHARING:
Plan to Share IPD: Yes
The researcher undertaking the qualitative interviews will get access to the patient identifier for those who have consented to take part in the interview so that they can access their contact details from the hospital record.
Supporting Information: CSR
Time Frame: The study findings will be submitted to a peer review journal within 6 months of study completion.
Access Criteria: This will likely be an open source journal